CLINICAL TRIAL: NCT06680882
Title: The Second Hospital Affiliated Anhui University of Chinese Medicine
Brief Title: The Effect of Non-invasive Auricular Acupoint Stimulation on Slow Transmission Constipation
Acronym: AAS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Heng Deng, The Second hospital affiliated Anhui University of Chinese Medicine, The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AH2022056; No. 2023AH050848 (Other Grant/Funding Number: Scientific Research Project of Colleges and Universities of Anhui Province)
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Slow Transmission Constipation
Keywords: slow transmission constipation

STUDY DESIGN:
Intervention Model Description: slow transmission constipation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): The study group, comprising 30 individuals, received a combination therapy of non-invasive auricular acupoint stimulation and prucapride
  Interventions: Other: Auricular Acupoint Stimulation +prucapride
- control group (Other): also consisting of 30 patients, was administered prucapride as a monotherapy.
  Interventions: Drug: prucapride

INTERVENTIONS:
Other: Auricular Acupoint Stimulation +prucapride — The study group, comprising 30 individuals, received a combination therapy of non-invasive auricular acupoint stimulation and prucapride
  Arms: study group
Drug: prucapride — was administered prucapride as a monotherapy
  Arms: control group

SUMMARY:
Objective To examine the therapeutic effect and safety of non-invasive auricular acupoint stimulation application on patients with slow transmission constipation.

Methods In a randomized clinical trial, 60 patients diagnosed with slow transit constipation (STC), ranging in age from 40 to 75 years, were allocated into two distinct cohorts: a study group and a control group. The study group, comprising 30 individuals, received a combination therapy of non-invasive auricular acupoint stimulation and prucapride, while the control group, also consisting of 30 patients, was administered prucapride as a monotherapy. To assess the efficacy of the interventions, various parameters were monitored, including serum levels of Neuropeptide Y (NPY), nitric oxide (NO), fecal water content, and gastrointestinal (GI) transit. The comparative therapeutic outcomes were determined by calculating symptom scores.

ELIGIBILITY:
Inclusion Criteria: ① Conformity to the diagnostic benchmarks for STC as delineated in the Rome IV criteria; ② Absence of ingestion of any medication influencing gastrointestinal motility within the preceding three months; ③ Provision of informed consent after a comprehensive understanding of the study's objectives; ④ An age range of 40 to 75 years.

-

Exclusion Criteria: ① Withdrawal from the therapeutic regimen; ② Auricle or ear canal pathologies; ③ Organic defecation disorder; ④ Pregnant or lactating.

-

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-07 (Estimated); Primary Completion 2024-11-07 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
overall efficacy rate | From enrollment to the end of treatment at one week
  Symptoms were assessed both one week prior to and one week following treatment. The defecation time (scored as follows: 0 for ≤5 minutes; 1 for >5 to ≤15 minutes; 2 for >15 to ≤25 minutes; and 3 for >25 minutes) and the inter defecation interval (scored as the number of hours divided by 24) were recorded. The efficacy index was calculated using the formula: [(pretreatment score - posttreatment score)/ pretreatment score] × 100%.

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial, only IPD used in the results publication